CLINICAL TRIAL: NCT06625021
Title: The Effect of Chiropractic and Different Physiotherapy Applications on Wrist Proprioception and Grip Strength in People With Mechanical Neck Pain
Brief Title: Effects of Chiropractic and Exercise on Wrist Proprioception and Grip Strength in Individuals With Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Ersin Cozvelioglu, Principal Investigator, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01- Chiropractic.vs.exercise
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Neck Pain
Keywords: Chiropractic Manipulation; Grip Strength; Neck Pain of Mechanical Origin; Rehabilitation Exercise; Proprioception
MeSH Terms: conditions — Neck Pain | interventions — Manipulation, Chiropractic

STUDY DESIGN:
Intervention Model Description: 48 individuals diagnosed with mechanical neck pain were included in the study. The 48 individuals were randomly divided into 4 groups via the Randomizer.org website.
  * The first group is the control group(n=12); transcutaneous electrical nerve stimulation, ultrasound and appropriate neck exercises are planned to be applied every day for 4 weeks.
  * The second group is the chiropractic group(n=12) and will be applied twice a week for 3 weeks by me, a Bahcesehir University Chiropractic Masters graduate, targeting the lower cervicals.
  * Classic hand-wrist exercises group(n=12) such as range of motion, stretching and strengthening were applied to the third group in all directions of the wrist.
  * In the fourth group, proprioceptive exercises group(n=12) such as joint approximation, traction and mobilization, similar to the classic hand-wrist exercise group, will be performed every day for 4 weeks.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Experimental): -The first group is the control group (n=12); Transcutaneous electrical nerve stimulation, ultrasound and appropriate neck exercises are planned to be applied every day for 4 weeks.
  Interventions: Procedure: Exercises to be done for neck pain of mechanical origin
- Chiropractic Group (Active Comparator): -The second group is the chiropractic group and will be applied twice a week for 3 weeks by me, a Bahcesehir University Chiropractic Masters graduate (2017), targeting the lower cervicals.
  Interventions: Procedure: Chiropractic manipulation; Procedure: Exercises to be done for neck pain of mechanical origin
- Classic Hand-Wrist Exercises Group (Active Comparator): -Classic hand-wrist exercises such as range of motion, stretching and strengthening were applied to the third group in all directions of the wrist.
  Interventions: Procedure: Exercises to be done for neck pain of mechanical origin; Procedure: Classic Hand-Wrist Exercises
- Proprioceptive Exercises Group (Active Comparator): -In the fourth group, proprioceptive exercises such as joint approximation, traction and mobilization, similar to the classic hand-wrist exercise group, will be performed every day for 4 weeks.
  Interventions: Procedure: Exercises to be done for neck pain of mechanical origin; Procedure: Proprioceptive exercise group

INTERVENTIONS:
Procedure: Chiropractic manipulation — Chiropractic manipulation: Lower cervical chiropractic manipulation is a technique used to increase mobility and relieve pain in the lower vertebrae of the neck. However, such procedures should only be performed by trained chiropractors; if done incorrectly, they can lead to serious problems. The patient should be placed in a comfortable position. The supine or side-lying position is usually preferred. Contact is established with the transverse processes of the lower cervical vertebrae. High-velocity, Low-amplitude thrust is applied within anatomical limits.
  As a graduate of Bahcesehir University Chiropractic Masters Degree, I applied chiropractic twice a week for 3 weeks.
  Arms: Chiropractic Group
Procedure: Exercises to be done for neck pain of mechanical origin — Conservative treatment, which is frequently used in the treatment of mechanical neck pain, was planned. A warm-up period was defined with stretching exercises in all areas of neck movement. Again, isometric exercise should be 10 seconds in all directions. In addition to neck and shoulder mobility exercises, neck region posture exercises were included. It was planned to do these exercises for 4 weeks, 5 days a week, in all 4 groups.
Procedure: Classic Hand-Wrist Exercises — The participants of this group will be subjected to wrist range of motion (ROM), stretching and strengthening exercises. Measurements will be made in all axes of motion of the wrist, which are extension, flexion, ulnar and radial deviation. ROM exercises and stretching exercises were applied passively to all axes of motion within anatomical limits. At the last angles of the movement, the individual was forced and stretched without causing discomfort and waited at the last angles for a short time. Stretching exercises were performed five times for each movement. Strengthening exercises for all axes of movement of the wrist will be performed using dumbbells weighing 1 and 2 kilograms and an exercise band suitable for the persons endurance and strength. In exercises performed with dumbbells, all movements of the wrist will be performed against gravity. All applications were applied to the classical hand-wrist exercise group for at least half an hour every day for 4 weeks.
  Arms: Classic Hand-Wrist Exercises Group
Procedure: Proprioceptive exercise group — Similar to the classical wrist exercise group, the participants in this group were applied joint range of motion, stretching and strengthening exercises as well as proprioceptive exercises such as joint approximation, traction and mobilization. In addition to all axes of motion of the wrist, active and passive stretching exercises were applied to the forearm flexor and extensor muscles five times each. The resistance and repetition number were gradually increased according to the wrist strength and endurance of the individuals to at least 10 repetitions. Repetitive contraction and rhythmic stabilization techniques were used from proprioceptive neuromuscular facilitation methods. Joint approximation technique and taping of forearm flexor and extensor muscles were used to increase the level of contraction and stimulation of joint receptors. External stabilization and perturbation exercises were performed with an exercise ball against the wall at different angles of the upper extremity.
  Arms: Proprioceptive Exercises Group

SUMMARY:
The aim of this study is to compare the effectiveness of chiropractic and different physiotherapy applications on bilateral hand grip strength, grip sensitivity, two-point separation and joint position sense in individuals with mechanical neck pain (NPMO). It is known that the decrease in grip strength and hand functions, especially with increasing age, causes disability in daily life activities and even death. The planned study aims to improve hand functions in individuals with NPMO.

48 individuals diagnosed with mechanical neck pain were included in the study. The 48 individuals were randomly divided into 4 groups via the Randomizer.org website.

* The first group is the control group (n=12); transcutaneous electric nerve stimulation, ultrasound and appropriate neck exercises are planned to be applied every day for 4 weeks.
* The second group is the chiropractic group and will be applied twice a week for 3 weeks by me, a Bahcesehir University Chiropractic Masters graduate (2017), targeting the lower cervicals.
* Classic hand-wrist exercises such as ROM, stretching and strengthening were applied to the third group in all directions of the wrist.
* In the fourth group, proprioceptive exercises such as joint approximation, traction and mobilization, similar to the classic hand-wrist exercise group, will be performed every day for 4 weeks.

The researcher will compare the effects of chiropractic and other physiotherapy techniques with the control group. Measurements will be repeated 4 weeks after the end of the treatment to measure whether the effects after the treatment continue. As a result of the evaluations recorded in a total of 8 weeks, statistical analyses will be performed first for the changes within the four groups and then for the changes between the groups.

The basic questions it aims to answer are as follows:

1. Is there a difference between the control group and chiropractic application, classic hand-wrist exercises and proprioceptive exercises in terms of the effects on grip strength, grip sensitivity, joint position sense and two-point discrimination test in individuals with NPMO?
2. Is there an improvement in the pain levels and functional disabilities of the participants?
3. Are the short-term results of the treatments sufficient?

DETAILED DESCRIPTION:
The brains primary means of survival is to receive and interpret sensory input. Therefore, it needs functional afferent inputs that can adapt to changing internal and external environmental conditions and update themselves. Most of this occurs through joint-based proprioceptive and muscle spindle information coming to the spinal code. The spinal cord is not only a center responsible for transmitting sensations coming to the dorsal horn to the brain, but also responsible for regulating these sensations. Due to the continuous afferent firing of the neck pain of mechanical origin (NPMO), the sensory-motor integration of the spinal cord decreases. When the afferent input of the spinal cord changes, it will not be possible to perceive correctly what is happening in the relevant region. It can be said that this situation affects itself in a cycle by changing sensory processing, sensory filtering and sensory integration. It can also cause the vertebral column to be exposed to microtrauma. With the decrease in the firing of the existing altered sensory inputs, joint position sense and motor control reach an optimum level, and increases have been observed in the regulation of developmental and physiological processes, especially in postural strength and upper extremity muscle strength. It is aimed to examine the relationship between the improvement of proprioceptive input with treatment methods and the elimination of abnormal motor control and abnormal neuronal processing with improved proprioceptive input. In this context, it was planned to evaluate the superiority of chiropractic, classical hand-wrist exercises and proprioceptive exercises against each other and against the control group in individuals with NPMO by applying grip strength, grip sensitivity, wrist joint position sense and 2-point discrimination test. It was planned to use visual analog scale and neck pain and disability score to assess pain in NPMO and Copenhagen neck functional disability scale to assess functionality.

With this study;

1. Ensuring normal integration in individuals with NPMO,
2. Ensuring sensory-motor integration by keeping the internal and external body schemas of the brain working healthily and up-to-date,
3. Increasing the pain and disability in daily activities and increasing the functionality by improving the strength and proprioception parameters of the hand and wrist,
4. Obtaining information about the general health of the individual by evaluating the grip strength and proprioception,
5. Providing higher quality health services with the findings obtained,
6. Guiding patients with evidence during the treatment process,
7. Providing the most appropriate treatment to patients is aimed.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with mechanical neck pain
* Presence of mechanical neck pain that has been ongoing for at least 14 days
* Newly starting conservative treatment for mechanical neck pain
* Age range 18-50 Exclusion criteria for the study

Exclusion Criteria:

* Individuals wanting to withdraw from the study
* Not signing the informed consent form
* Using painkillers for neck pain of mechanical origin pain during the application period
* Presence of upper extremity trauma that may affect grip strength and proprioceptive sense in the last 3 months
* Vertebrobasilar artery insufficiency
* Presence of mental retardation and/or inability to communicate
* Having undergone surgery in the cervical region
* Presence of neck pain of neurological origin such as stenosis and herniation of cervical segments
* Presence of sensory deficit in the hand

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2023-01-21 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | The first measurements will be taken before treatment. The second measurements are planned to be taken at the end of treatment, 4 weeks after the start. The third measurements will be taken 8 weeks after the start to evaluate the early effects.
  Visual Analog Scale (VAS) is used to make some values numerically measurable. In order to measure the pain values of all participants subjectively, it is possible to evaluate their pain on a horizontal plane scale of 0-10 centimeters (cm) or 0-100 millimeters (mm). They were asked to mark the values of the pain they felt, with 0 mm indicating no pain and 10 cm or 100 mm indicating the maximum possible pain. The participants were given definitions of the two extreme parts of the VAS and the patients were asked to indicate where their pain was appropriate by making a mark, drawing a line or verbally and recorded in centimeters. The VAS values of the individuals participating in the study were recorded before the treatment, after the treatment and 4 weeks after the end of the treatment, while resting and during activity.
Neck pain and disability scale | The first measurements will be taken before treatment. The second measurements are planned to be taken at the end of treatment, 4 weeks after the start. The third measurements will be taken 8 weeks after the start to evaluate the early effects.
  The validity and reliability of the adaptation of the Neck Pain and Disability Scale (NPDS) to Turkish has been proven. In addition to the evaluation of pain, it examines the effects of pain intensity on social, functional, emotional, daily life activities, recreational and occupational factors. Thus, the 29 effects of neck pain on functionality, quality of life and disability are measured. The NPDS, which consists of 20 items, uses a score between 0 and 5. While the scores of each question can be added up to a value between 0 and 100, the higher the total scores, the more severe the pain and the worse the pain is affected.
Copenhagen neck functional disability scale | The first measurements will be taken before treatment. The second measurements are planned to be taken at the end of treatment, 4 weeks after the start. The third measurements will be taken 8 weeks after the start to evaluate the early effects.
  The Copenhagen neck functional disability scale is used to measure neck functionality in the presence of neck pain. It is a scale consisting of 15 items that investigates individuals' self-care, sleep status, disability in daily life and social life impact. It measures pain intensity, independence in daily life or disability, future anxiety of pain, social impact and impact during recreational activities. For the first 5 questions, the Yes answer is (0) points, the Occasional answer = (1) points, the No answer is (2) points. For the other questions, the Yes answer is (2) points, the Occasional answer is (1) points, and the No answer is (0) points. Scoring of the scale; While the total score is calculated between 0 and 30 points, the higher the total score, the higher the minimal disability level, and the lower the total score, the lower the minimal disability.
Grip strength | The first measurements will be taken before treatment. The second measurements are planned to be taken at the end of treatment, 4 weeks after the start. The third measurements will be taken 8 weeks after the start to evaluate the early effects.
  A Baseline brand hand dynamometer, which is a frequently used device for measuring hand grip strength, was used. The measurements were made with the participants sitting with their arms next to their bodies, 90° elbow flexion, and the forearm in neutral position, and the wrist in 0 to 30° extension for maximal grip strength. The measurements were made bilaterally, with short rest periods, in three measurements. The arithmetic average of the 3 measurements measured bilaterally was taken for evaluation.
Grip force sensitivity | The first measurements will be taken before treatment. The second measurements are planned to be taken at the end of treatment, 4 weeks after the start. The third measurements will be taken 8 weeks after the start to evaluate the early effects.
  In order to evaluate the sensitivity of grip force or in other words, the sensitivity of grip pressure, the Baseline brand Pneumatic Bulb Dynamometer device was used. Pneumatic devices have an air-filled bulb-like shape and provide the measurement of grip force. Individuals grip strengths were measured with the Baseline Pneumatic Bulb Dynamometer device. By targeting half of the maximum grip force, the device indicator was shown to the individuals and they were asked to apply 50% of their maximal grip force, keep it in their memory and repeat it. After a few repetitions, the targeted force was asked to be repeated without showing the device screen and the absolute value of the difference was noted. The evaluation was repeated 3 times and recorded as grip force sensitivity error. A few minutes of rest were given for situations such as fatigue and loss of motivation.
Joint position sense | The first measurements will be taken before treatment. The second measurements are planned to be taken at the end of treatment, 4 weeks after the start. The third measurements will be taken 8 weeks after the start to evaluate the early effects.
  In the evaluation of range of motion(ROM) of the wrist, the recorded angles were grouped as actively repeated outside the visual field. All movement axes of the wrist were used for measurement. The target angle for extension and flexion movements of the wrist was defined as 30°, and ulnar and radial deviation angles were defined as 15° and 10°, respectively. ROM was evaluated three times in all movement axes and desired positions of the wrist, and the average of these 3 values was recorded as wrist ROM margin of error.

CONTACTS AND LOCATIONS:
Overall Officials: Ersin COZVELIOGLU, Ph.D, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaras Sutcu Imam University Health Practice and Research Hospital, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No